CLINICAL TRIAL: NCT05247918
Title: OBDIPHY (OBesity DIgital-PHYsical Care Study) - Effects of Digi-physical Care for Families
Brief Title: OBDIPHY (OBesity DIgital-PHYsical Care Study)
Acronym: OBDIPHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Region Skane (Other); Vastra Gotaland Region (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 276515
Record Dates: First submitted 2021-12-07; First posted 2022-02-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Pediatric Obesity; Obesity; Adolescent Obesity; Lifestyle Risk Reduction; Metabolic Syndrome; Weight Loss
MeSH Terms: conditions — Pediatric Obesity; Obesity; Risk Reduction Behavior; Metabolic Syndrome; Weight Loss | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Multicenter prospective randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital-physical care group (Experimental): Combination of digital and physical care.
  Interventions: Behavioral: Digital-physical care
- Treatment as usual. (Active Comparator): Treatment as usual in accordance with national guidelines.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Digital-physical care — Patients will get access to a digital communication platform. Two in person session and two digital contacts per year with possibility to chat with caregivers in between.
  Arms: Digital-physical care group
Behavioral: Treatment as usual — Four in person session at the center in a year.
  Arms: Treatment as usual.

SUMMARY:
This is a prospective randomized controlled multicentre non-inferiority trial. The aim of this study to evaluate digi-physical care compared to regular physical/in person care and investigate if digi-physical care can be an equal or even better treatment alternative among families with children or adolescents living with obesity in Sweden. The study participants will either get treatment as usual or treatment as usual combined with digi-physical solution. The digi-physical solution includes thar half of the session is digital and they get an app where they can self-monitoring health data, have an overview over they treatment plan and easy communicate with theirs caregivers.

DETAILED DESCRIPTION:
This study is multi centre in three different county council in southwest of Sweden which include children and adolescents in the age of 10-16 year. The study participants will either get treatment as usual, which includes four in person session with healthcare professionals as doctor, nurse or dietitian (the control group) or treatment as usual combined with digi-physical solution (intervention group). The intervention group will beyond treatment as usual get a digital communication platform (including an app) where the patient has a good overview of their treatment plan, can report self-monitored health data as daily steps and weight once a week and monitor the daily work with their selected health goal. Everything in the app is individually tailored together with the patient. The patient with digi-physical care will also have assess to a chat for communication with their caregivers. The app has a high degree of authentication and classified as a journal system. Half of yearly treatment as usual sessions will be digital for the intervention group.

The digi-physical method of treatment is developed and based on the desire from the patient association HOBS (hälsa oberoende av storlek). In parts of Sweden people have long distance to the clinic which makes it difficult to be present at the treatment in-clinic sessions and the families loses many hours away from school and work. The null hypothesis is that digi-physical care will have a positive effect on BMI SDS, however inferior to treatment as usual.

In addition to evaluate that this new treatment alternative is safe will also ISO-BMI, weight development and metabolic risk factors be evaluated. The study does not include any extra blood samples or visits to the clinic thus everything is collected according to regular care programs. To evaluate the food intake and possible changes there will be three 24-h recalls, combined with riksmaten flex, performed. There will also be questions about their physical activity and a survey (PEDS-QL) for mental health. For a few volunteered patient families, approximate 15-20, will participate in semi-structured deep interviews.

ELIGIBILITY:
Inclusion Criteria:

* ISO-BMI 30 or above.

Exclusion Criteria:

* Lack of Swedish skills
* Patients potential for obesity surgery
* Patient with obesity syndrome

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in BMI standard deviation score at month 12. | Baseline and month 12.
  The BMI standard-deviation score is a measure of the number of standard deviations from the population mean BMI (weight divided by height squared), matched for age and sex.

SECONDARY OUTCOMES:
Change from baseline in BMI standard deviation score at month 6. | Baseline and month 6.
  The BMI standard-deviation score is a measure of the number of standard deviations from the population mean BMI (weight divided by height squared), matched for age and sex.
Change from baseline in BMI standard deviation score at month 18. | Baseline and month 18
  The BMI standard-deviation score is a measure of the number of standard deviations from the population mean BMI (weight divided by height squared), matched for age and sex.
Change from baseline in weight at month 3. | Baseline and month 3.
  Weight in kilogram measure in clinic at the hospital scales from TANITA or self monitored at home on a Beurer BF 850 scale.
Change from baseline in weight at month 6. | Baseline and month 6.
  Weight in kilogram measure in clinic at the hospital scales from TANITA or self monitored at home on a Beurer BF 850 scale.
Change from baseline in weight at month 9. | Baseline and month 9..
  Weight in kilogram measure in clinic at the hospital scales from TANITA or self monitored at home on a Beurer BF 850 scale.
Change from baseline in weight at month 12. | Baseline and month 12.
  Weight in kilogram measure in clinic at the hospital scales from TANITA or self monitored at home on a Beurer BF 850 scale.
Change from baseline in weight at month 18. | Baseline and month 18.
  Weight in kilogram measure in clinic at the hospital scales from TANITA or self monitored at home on a Beurer BF 850 scale.
Change from baseline in waist circumference at 6 and 12 month. | Baseline and month 6 and 12.
  Waist circumference measure in cm with measuring tape.
Change from baseline in waist circumference at 6 month. | Baseline and month 6.
  Waist circumference measure in cm with measuring tape.
Change from baseline in blood pressure at12 month. | Baseline and month 12.
  Bloodpressure in mm Hg, measured in right arm while sitting down after 5 minits of rest. It will be measured three times and then the mean of the two last measure will be calculated and reported.
Change from baseline in fasting insulin at 12 month. | Baseline and month 12.
  Fasting insulin from blood sample measured in mU/L. Analyzed according to standard routine.
Change from baseline in fasting glucose at 12 month. | Baseline and month 12.
  Fasting glucose from blood sample measured in mmol/L. Analyzed according to standard routine.
Change from baseline in HbA1c at 12 month. | Baseline and month 12.
  HbA1c from blood sample measured in mmol/L. Analyzed according to standard routine.
Change from baseline in lever enzymes, ASAT, at 12 month. | Baseline and month 12.
  ASAT from blood sample measured in µkat/L. Analyzed according to standard routine.
Change from baseline in lever enzymes, ALAT, at 12 month. | Baseline and month 12.
  ALAT from blood sample measured in µkat/L. Analyzed according to standard routine.
Change from baseline in triglyceride at 12 month. | Baseline and month 12.
  Triglyceride from blood sample measured in mmol/L. Analyzed according to standard routine.
Change from baseline in cholesterol at 12 month. | Baseline and month 12.
  Cholesterol from blood sample measured in mmol/L. Analyzed according to standard routine.
Change from baseline in blood lipid, LDL, at 12 month. | Baseline and month 12.
  LDL from blood sample measured in mmol/L. Analyzed according to standard routine.
Change from baseline in blood lipid, HDL, at 12 month. | Baseline and month 12.
  HDL from blood sample measured in mmol/L. Analyzed according to standard routine.
Change from baseline in food intake according to Riksmaten Flex and 24-hour recalls in 12 month. | Baseline and month 12.
  RiksmatenFlex and 24-hour recalls is a validated survey about food habits combined with three 24-hour interviews, where food intake the last 24 h are reported.
Change from baseline in amount of steps per day according to activity watch at week 52. | Baseline (week 1) and 52.
  Amount of daily steps will be self-monitored with a sportsbuddy veryfit activity watch and then selfreported in to the study app. The mean of one weeks step will be colected at week 1, 26 and 52.
Change from baseline in amount of steps per day according to activity watch at week 26. | Baseline (week 1) and week 26.
  Amount of daily steps will be self-monitored with a sportsbuddy veryfit activity watch and then selfreported in to the study app. The mean of one weeks step will be collected at week 1, 26 and 52.
Change from baseline in health-related quality of life according to PEDS-QL at 12 month | Baseline and month 12.
  PEDS-QL is a valid questionaire for evaluating health-related quality of life used by the Swedish childhood obesity treatment register (BORIS). The child will answer if they never, almost never, sometimes, often or always has experience diffrent issues conserning their health.
Change from baseline in daily well-being on a 10 point VAS-scale at week 26. | Baseline (week 1), and week 26.
  Daily self reported well-being via a VAS-scale from 1-10 (1=worst feeling, 10=best feeling). The mean of one week reported data will be collected at week 1, 26 and 52.
Change from baseline in daily well-being on a 10 point VAS-scale at week 52. | Baseline (week 1) and 52.
  Daily self reported well-being via a VAS-scale from 1-10 (1=worst feeling, 10=best feeling). The mean of one week reported data will be collected at week 1, 26 and 52.
Thoughts on implementation from caregivers after a 12-month digital-physical care. | At month 12
  Survey about caregivers experience through implementation of digital care. Few easy questions about positive and negative aspects.
Thoughts on implementation from patients after a 12-month digital-physical care. | At month 12
  Survey about patient experience through implementation of digital care. Few easy questions about positive and negative aspects and how they used the app.
Semi-structured interviews for a deeper insight in the qualitative aspects concerning digital care. | At month 12.
  Semi-structured interviews with 15-20 of the patient families inte the intervention group. The interview will proceed from open answer questions with the possibility to expand answers.

OTHER OUTCOMES:
Report digital selfmonitored health data. | At 3 month.
  Evaluate the precentage of typ 2 diabetes patientens that reported self-monitored health data by the digital communication platform.

CONTACTS AND LOCATIONS:
Overall Officials: Josefin Roswall, Study Chair — Region Halland
Locations (5):
- Sweden (5):
  - Regionalt obesitascentrum, Gothenburg
  - Barnkliniken Halland, Halmstad
  - Barnkliniken Halland, Kungsbacka
  - Överviktenheten Barn, Malmo
  - Barnkliniken Halland, Varberg

IPD SHARING:
Plan to Share IPD: No